CLINICAL TRIAL: NCT06394375
Title: Effectiveness of Opioid Free Anesthesia Using Dexmedetomidine Inhibiting Nociception in Abdominal Laparoscopic Surgery
Brief Title: Opioid Free Anesthesia in Abdominal Laparoscopic Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aida Rosita Tantri, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IndonesiaU23061029
Record Dates: First submitted 2024-04-20; First posted 2024-05-01 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Laparoscopic Surgery; Abdominal Surgery
Keywords: Abdominal surgery; Laparoscopic surgery; Dexmedetomidine; Opioid free anesthesia
MeSH Terms: interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Intervention Model Description: Participants are randomized into two groups for control (opioid balanced anesthesia) or intervention (opioid free anesthesia)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid free anesthesia (Experimental): Patients in this group are given a combination of Dexmedetomidine, Lidocaine, Propofol, Sevoflurane, Rocuronium for induction and maintenance of general anesthesia. They are given rescue analgesia (fentanyl) when required, and Ephedrine as needed.
  Patients were monitored using standard ASA monitoring and Connox.
  Post operative pain score was assessed with NRS
  Interventions: Drug: Dexmedetomidine
- Opioid balanced anesthesia (Active Comparator): Patients in this group are given a combination of Opioid (Fentanyl), Lidocaine, Propofol, Sevoflurane, Rocuronium for induction and maintenance of general anesthesia. They are given Ephedrine as needed.
  Patients were monitored using standard ASA monitoring and Connox.
  Post operative pain score was assessed with NRS
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Dexmedetomidine — OFA
  Arms: Opioid free anesthesia
Drug: Fentanyl — Given as analgesia in opioid balanced anesthesia (control) group
  Arms: Opioid balanced anesthesia

SUMMARY:
Effectiveness of opioid free anesthesia using Dexmedetomidine to inhibit nociception in abdominal laparoscopic surgery

DETAILED DESCRIPTION:
Abdominal laparoscopic surgery is one of the most common procedures worldwide, commonly facilitated with opioid balanced anesthesia or regional anesthesia. Despite being a controversy, there are issues that suggest opioid to have an influence in tumor recurrence. The investigators performed general anesthesia without opioid in laparoscopic abdominal surgery, and compared the hemodynamic instability, total consumption of fentanyl rescue, qNOX score, Ephedrine intraoperative, and Numerical Rating Scale.

ELIGIBILITY:
Inclusion criteria

* Patients undergoing abdominal laparoscopic surgery (digestive, urologic, gynecologic surgery) with general anesthesia
* BMI <= 30 kg/m2
* Assessed with ASA 1-3
* Willing to participate in this study

Exclusion Criteria:

* Allergy to dexmedetomidine
* Heart rate < 60 or systolic blood pressure <100 mmHg
* Severe cardiovascular, uncontrolled hypertension (stage 2) or hepatic or renal disorder
* Sepsis
* Pregnancy
* Difficult airway

Drop out Criteria:

* Intraoperative emergency
* Convert to open laparatomy
* Decided to withdraw from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Intraoperative
  blood pressure, both systolic and diastolic measured with non invasive blood pressure monitoring
Heart rate | Intraoperative
  Heart rate

SECONDARY OUTCOMES:
Total consumption of Opioid | Intraoperative
  Total consumption of fentanyl as rescue analgesia in mcg
quantium nociception index (qNOX) | Intraoperative
  qNox score is measured at specific time points, available from Conox monitor measurement since the start of the procedure. Higher value indicates more nociception experienced by the patient (0-100)
Ephedrine | intraoperative
  Total consumption of ephedrine to increase heart rate and blood pressure in mg
Pain score | 24 hour
  Numerical rating scale 0-10 is used to quantify pain score postoperatively, with higher value indicating more pain experienced by the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia